CLINICAL TRIAL: NCT01183572
Title: Trial of Pre-Pregnancy Supplements
Acronym: TOPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Ifakara Health Institute (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Chair, Department of Global Health and Population, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0055/07
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Anemia
Keywords: multivitamins; folate; iron; periconception
MeSH Terms: conditions — Anemia | interventions — Geritol; Folic Acid; Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Folic Acid and Iron (Active Comparator): 0.4mg of folic acid and 30 mg elemental iron taken daily for 6 months
  Interventions: Dietary Supplement: Folic Acid and Iron
- Folic Acid (Placebo Comparator): 0.4mg of folic acid taken daily for 6 months
  Interventions: Dietary Supplement: Folic Acid
- Multivitamins, Folic Acid, and Iron (Active Comparator): A multivitamin and micronutrient supplement that constitutes 1 RDA of Vitamins A (2500 IU), B1 (1.4 mg), B2 (1.4 mg), B6 (1.9 mg), B12 (2.6 ug), niacin (18 mg), C (70 mg), E (10 mg), and folic acid (0.4 mg)along with 30 mg of elemental iron taken daily for 6 months.
  Interventions: Dietary Supplement: Multivitamins, Folic Acid, and Iron

INTERVENTIONS:
Dietary Supplement: Multivitamins, Folic Acid, and Iron — Daily oral dose containing 2500 IU Vitamin A, 1.4 mg Vitamin B1, 1.4 mg Vitamin B2, 2.6 mg Vitamin B12, 1.9 mg Vitamin B6, 18 mg Niacin, 70 mg Vitamin C, 14.9 IU Vitamin E, 30 mg elemental iron, 0.4 mg folic acid
  Arms: Multivitamins, Folic Acid, and Iron
Dietary Supplement: Folic Acid and Iron — Daily oral dose of 30 mg elemental iron, 0.4 mg folic acid
  Arms: Folic Acid and Iron
Dietary Supplement: Folic Acid — Daily oral dose of 0.4 mg folic acid
  Arms: Folic Acid

SUMMARY:
The purpose of this study is to determine whether daily oral supplements of multivitamins (including vitamins B-complex, C and E) along with Iron and folic acid given to non-pregnant women results in lower prevalence of anemia in preparation for pregnancy when compared to daily iron and folic acid supplements or folic acid alone.

DETAILED DESCRIPTION:
Globally, more than half a million women die from pregnancy or childbirth-related complications, most of them in developing countries. The global community committed to reducing the maternal mortality ratio by three quarters between 1990 and 2015 (MDG5). Women die from a range of complications in pregnancy, childbirth or the postpartum period. 80% of maternal deaths are due to severe bleeding (mostly bleeding postpartum), infections, hypertensive disorders in pregnancy and obstructed labor. Additionally, low birth weight and neonatal mortality are common problems in developing countries. The benefit of periconceptual folate on preventing congenital anomalies has been established in randomized trials; however, the role of other nutrients needs to be examined further. Anemia is strongly associated with adverse perinatal outcomes including maternal mortality and low birthweight.

ELIGIBILITY:
Inclusion Criteria:

1. Girls aged > =15 years and <= 29 years
2. Have not missed a menstrual period during recruitment (no amenorrhea)
3. Has not been pregnant or given birth within the last 6 months
4. Intend to stay in the study area for at least 6 months after enrollment
5. Have provided written informed consent

Exclusion Criteria:

1. Amenorrhea or confirmed pregnancy at screening or enrollment.
2. Has given birth within 6 months
3. Already taking long-term vitamin supplementation.
4. Any severe illness requiring hospitalization at screening or enrollment (women who have been deemed to have recovered will be eligible once they return home).

Ages: 15 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 802 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Anemia | 6 months following the start of the intervention
  Anemia will be defined as hemoglobin < 12gm/dL at 6 months of intervention. Hemoglobin concentration will also be analyzed as a continuous outcome.

SECONDARY OUTCOMES:
Weight Gain during intervention | 6 months following the start of the intervention
  Weight gain during intervention will be defined as the difference in weight between weight at randomization and weight at 6 months of intervention.
Mid Upper Arm Circumference | 6 months following the start of the intervention
Peripheral malaria parasitemia | 6 months following the start of the intervention
  Peripheral malaria parasitemia will be defined as fever in the past 72 hours with any malaria parasitemia in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MD, DrPH, Principal Investigator — Harvard School of Public Health (HSPH); Honorati M Masanja, PhD, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute, Rufiji, Tanzania

REFERENCES:
- [Derived] Gunaratna NS, Masanja H, Mrema S, Levira F, Spiegelman D, Hertzmark E, Saronga N, Irema K, Shuma M, Elisaria E, Fawzi W. Multivitamin and iron supplementation to prevent periconceptional anemia in rural tanzanian women: a randomized, controlled trial. PLoS One. 2015 Apr 23;10(4):e0121552. doi: 10.1371/journal.pone.0121552. eCollection 2015. PMID 25905863